CLINICAL TRIAL: NCT07046299
Title: Safety and Efficacy of Endovascular Therapy for Acute Basilar Artery Occlusion With Large Core Infarct: A Prospective, Multicenter, Randomized, Open-Label Controlled Trial
Brief Title: Basilar Artery Occlusion Chinese Endovascular Trial in Patients With Large Core Infarct
Acronym: BAOCHE3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAOCHE3
Record Dates: First submitted 2025-06-18; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Basilar Artery Occlusion; Ischemic Stroke; Large Core Infarct
Keywords: Endovascular Therapy; Large Core Infarct; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Therapy Plus Best Medical Treatment (Experimental): Patients randomized to this arm will receive endovascular therapy (EVT) in addition to best medical treatment. EVT must be initiated within 24 hours of symptom onset and completed within 3 hours.The EVT strategy will be selected by the treating neurointerventionalist based on vascular findings. Allowed procedures include mechanical thrombectomy, intra-arterial thrombolysis, balloon angioplasty, stent implantation, or a combination of these.
  Interventions: Procedure: Endovascular Therapy Plus Best Medical Treatment
- Best Medical Treatment Alone (Active Comparator): Patients in this arm will receive best medical treatment alone in accordance with current stroke guidelines. No endovascular therapy will be performed.
  Interventions: Drug: Best Medical Treatment Alone

INTERVENTIONS:
Procedure: Endovascular Therapy Plus Best Medical Treatment — Participants assigned to the endovascular therapy arm will receive EVT in addition to best medical treatment. EVT must be initiated within 24 hours of symptom onset and completed within 3 hours of groin puncture. After evaluating vascular anatomy, neurointerventionalists will determine the most appropriate strategy based on the presence of proximal stenosis, occlusion morphology, and vessel tortuosity. Permitted interventions include mechanical thrombectomy, stent thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, balloon angioplasty, and stent implantation. The choice of treatment approach is left to the discretion of the treating physician, and combinations of techniques are allowed.
  Other Names: Mechanical Thrombectomy
  Arms: Endovascular Therapy Plus Best Medical Treatment
Drug: Best Medical Treatment Alone — Participants in this arm will receive best medical treatment and maximal supportive care according to current stroke guidelines, without the use of mechanical thrombectomy or any intra-arterial intervention.
  Arms: Best Medical Treatment Alone

SUMMARY:
This study evaluates the safety and efficacy of endovascular therapy for acute basilar artery occlusion with large core infarcts in a multicenter randomized trial.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, controlled trial evaluating endovascular therapy (EVT) for patients with acute basilar artery occlusion (BAO) and large core infarcts, defined by a pc-ASPECTS score of 3-5 on DWI or CT. Eligible participants aged 18-80 years and presenting within 24 hours of symptom onset will be randomly assigned in a 1:1 ratio to receive either EVT plus standard medical therapy or medical therapy alone. Randomization will be stratified by age, baseline NIHSS, and onset-to-treatment time. The primary outcome is the proportion of patients achieving functional independence (mRS 0-3) at 90 days. Secondary outcomes include neurological improvement, mRS distribution, quality of life, and 90-day all-cause mortality, and the incidence of symptomatic intracranial hemorrhage (sICH). This study aims to generate high-quality evidence to guide treatment strategies for patients with acute basilar artery occlusion and large core infarcts.

ELIGIBILITY:
Inclusion Criteria:

1. Posterior circulation acute ischemic stroke within 24 hours from symptom onset/last seen well.
2. Occlusion (TIMI 0-1) of the basilar artery or intracranial segments of both vertebral arteries (V4) as evidenced by CTA/MRA/DSA.
3. Patients with large core infarction in the posterior circulation, defined as a posterior circulation Acute Stroke Prognosis Early CT score (pc-ASPECTS) score of 3-5 on CT angiography source images or MR with diffusion-weighted imaging or non-contrast CT.
4. Age ≥18 and ≤80 years.
5. Baseline NIHSS score ≥6 at the time of randomization.
6. No significant pre-stroke functional disability (modified Rankin Scale, mRS ≤ 1).
7. Informed consent obtained from patient or acceptable patient surrogate.

Exclusion Criteria:

Clinical exclusion criteria:

1. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0.
2. Baseline platelet count < 50000/µL.
3. Baseline blood glucose of < 50mg/dL or >400mg/dL.
4. Severe, sustained hypertension (SBP > 220 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained below these levels using commonly used medications in China for these purposes (including iv antihypertensive drips), the patient can be enrolled.
5. Patients in whom baseline NIHSS can not be obtained by a neurologist or emergency physician prior to sedation or intubation.
6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS.
7. Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
8. History of life threatening allergy (more than rash) to contrast medium.
9. Patients with acute stroke within the first 48 hours after percutaneous cardiac, cerebrovascular interventions and major surgery .
10. Renal insufficiency with creatinine ≥ 3 mg/dL.
11. Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
12. Subject participating in a study involving an investigational drug or device that would impact this study.
13. Known diagnosis or clinical suspicion of cerebral vasculitis.
14. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
15. Unlikely to be available for 90 days follow-up (e.g. no fixed home address, visitor from overseas).

    Neuroimaging exclusion criteria:
16. Pons-midbrain-index of ≥ 4 on CT angiography source images or MR with diffusion-weighted imaging or non-contrast CT.
17. CT or MR evidence of hemorrhage (the presence of microbleeds on MRI is allowed).
18. Complete cerebellar infarct on CT or MRI with significant mass effect and compression of the fourth ventricle.
19. Complete bilateral thalamic infarction on CT or MRI.
20. Evidence of vertebral occlusion, high grade stenosis or arterial dissection in the extracranial or intracranial segment that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment.
21. Subjects with occlusions in both anterior and posterior circulation.
22. Evidence of intracranial tumor (except small meningioma).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Achieving mRS 0-3 at 90 Days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death]). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Dramatic early favorable response | 24 (-2/+12) hours
  Dramatic early favorable response as determined by an National Institute of Health stroke scale (NIHSS) of 0-2 or NIHSS improvement ≥ 8 points at 24 (-2/+12) hours.
Ordinal Shift analysis of mRS at 90 days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Dichotomized mRS score (0-2 versus 3-6 ) | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Proportion of Patients Achieving mRS 0-4 at 90 Days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Barthel Index | 90 days
  The Barthel Index ranges from a minimum of 0 to a maximum of 100, with higher scores indicating better outcomes.
Proportion of patients achieving favourable outcomes defined as mRS 0-3 at 6 months | 6 months
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Proportion of patients achieving favourable outcomes defined as mRS 0-3 at 12 months | 12 months
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Proportion of basilar artery recanalization | 24 hours (-2/+12 hours)
  Vessel recanalization at 24 hours (-2/+12 hours) in both treatment groups assessed by using Arterial Occlusive Lesion (AOL) grades

OTHER OUTCOMES:
Mortality | 90 days
Symptomatic intracranial hemorrhage | 24 (-2/+12) hours
Serious adverse events | 90 days, 12 months, through study completion ( average of 1 year)
  All serious adverse events during follow-up in all randomized patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.